CLINICAL TRIAL: NCT00149994
Title: DELTA Study Dutch Evaluation in Liver Transplantation To Assess the Efficacy of Cyclosporine A Microemulsion With C-2h Monitoring Versus Tacrolimus With Trough Monitoring in de Novo Liver Transplant Recipients
Brief Title: Cyclosporine A C-2h Monitoring Versus Tacrolimus C-0h Monitoring in de Novo Liver Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: COLO400ANL07
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Results first posted 2011-02-14 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2011-04

CONDITIONS: Liver Transplant
Keywords: Liver transplant, adults, C2 monitoring
MeSH Terms: interventions — Cyclosporine; Tacrolimus; Basiliximab; Methylprednisolone; Prednisone

ARMS (2):
- Cyclosporine A (Experimental): Cyclosporine A was given in a twice-daily schedule at 12-hour intervals. It was administered within the first 4 hours post-operatively (study day 1), at an initial dose of 10-15mg/kg/day in two doses, as close as possible to 15mg/kg/day. After the first oral administration, the dose of Cyclosporine A was adjusted to bring the sample taken 2 hours after oral dose (C-2h) level into the target range by Days 3-5 post-transplantation. C-2h target ranges post-transplantation: 0-3 months: range of 800-1200 ng/ml with midpoint of 1000 ng/ml; 4-6 months: range of 700-900 ng/ml with midpoint of 800 ng/ml; > 6 months: range of 500-700 ng/ml with midpoint of 600 ng/ml is recommended. During the course of the study, the dose of Cyclosporine A was adjusted as necessary to achieve and maintain the C-2h blood Cyclosporine A (CsA) concentrations within the target ranges.
  Interventions: Drug: Cyclosporine A; Drug: Basiliximab; Drug: Methylprednisolone; Drug: Prednisone
- Tacrolimus (Active Comparator): Tacrolimus was given on a twice-daily schedule at 12-hour intervals which had to be maintained throughout the study period. Tacrolimus was administered within the first 24 hrs postoperatively (Study Day 1) at an initial dose of 0.1-0.15 mg/kg/day in two divided oral doses either by mouth or via an enteral feeding tube until the patient can swallow. The initial dosing level was determined by the patient's overall post-operative condition. During the course of the study, the dose of tacrolimus was adjusted as necessary to achieve and maintain the pre-dose blood concentration (C-0h) (trough) tacrolimus concentrations. C-0h target ranges post-transplantation: 0-3 months: 10-15 ng/ml; 4-6 months: 5-10 ng/ml; > 6 months: range of 5-10 ng/ml is recommended.
  Interventions: Drug: Tacrolimus; Drug: Basiliximab; Drug: Methylprednisolone; Drug: Prednisone

INTERVENTIONS:
Drug: Cyclosporine A
  Arms: Cyclosporine A
Drug: Tacrolimus
  Arms: Tacrolimus
Drug: Basiliximab — Each patient was given two 20mg doses of Basiliximab as intravenous bolus injection at Day 0 and Day 4 post-transplant surgery.
Drug: Methylprednisolone — Methylprednisolone was given as an intravenous bolus of 500mg during transplant surgery
Drug: Prednisone — Post-operatively prednisone was tapered from an initial dose of 20mg/day to zero at 3 months or continued at 5-10mg if the indication for Orthotopic Liver Transplantation (OLTx) was of auto-immune nature.

SUMMARY:
The purpose of this study is to determine whether cyclosporine A (in a micro emulsion formulation) monitored by sample taken 2 hour after oral dose (C-2h) will show equivalent or superior efficacy compared to tacrolimus monitored by pre-dose blood concentration (C-0h). In addition this study will assess the safety and tolerability of a cyclosporine A regimen based on C-2h monitoring in comparison to the standard tacrolimus regimen.

ELIGIBILITY:
Inclusion Criteria:

* About to undergo a primary liver transplant (including living donor, non-heart beating donor and split liver).
* Age between 18 and 75 years.
* Expected to be able to receive the first oral dose of CNI within the first 24 hours post-transplantation (Tx)

Exclusion Criteria:

* This is a multi-organ transplant or if the patient has previously been transplanted with any other organ.
* Urine production is <200 ml within 12 hours after reperfusion of the graft
* Severe coexisting disease is present or if any unstable medical condition is present which could affect the study objectives.

Other protocol-defined exclusion criteria applied

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2002-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis, Basel, Switzerland

RESULTS

PARTICIPANT FLOW:
Groups:
- Cyclosporine A: Cyclosporine A was given twice-daily at 12-hour intervals. It was administered within the first 4 hours post-operatively (study day 1), at an initial dose of 10-15mg/kg/day in two doses. Cyclosporine A was adjusted to bring the 2 hour after oral dose (C-2h) level into the target range by Days 3-5 post-transplantation. The dose of Cyclosporine A was adjusted to achieve and maintain post transplantation C-2h levels 0- 3 months: 800- 1200 ng/mL, 4- 6 months: 700- 900 ng/mL and >6 months: 500- 700 ng/mL. Each participant was given two 20 mg doses of Basiliximab as intravenous bolus injection at Day 0 and Day 4 post-transplant surgery. Methylprednisolone was given as an intravenous bolus of 500 mg during transplant surgery. Post-operatively prednisone was tapered from an initial dose of 20 mg/day to zero at 3 months or continued at 5-10 mg if the indication for Orthotopic Liver Transplantation (OLTx) was of auto-immune nature.
- Tacrolimus: Tacrolimus was given twice-daily at 12-hour intervals. Tacrolimus was administered within the first 24 hrs post- operatively (Study Day 1) at an initial dose of 0.1-0.15 mg/kg/day in two divided oral doses either by mouth or via an enteral feeding tube until the participant can swallow. The initial dosing level was determined by the participants's overall post-operative condition. The dose of tacrolimus was adjusted to achieve and maintain the pre-dose C-Oh (trough) target ranges post-transplantation 0-3 months: 10-15 ng/ml; 4-6 months: 5-10 ng/ml and > 6 months: 5-10 ng/ml . Each participant was given two 20 mg doses of Basiliximab as intravenous bolus injection at Day 0 and Day 4 post-transplant surgery. Methylprednisolone was given as an intravenous bolus of 500 mg during transplant surgery. Post-operatively prednisone was tapered from an initial dose of 20 mg/day to zero at 3 months or continued at 5-10 mg if the indication for OLTx was of auto-immune in nature.
Period: Overall Study
Arm/Group | Cyclosporine A | Tacrolimus
Started | 85 ("Started" indicates Safety population.) | 86
Completed | 84 ("Completed" indicates intention to treat (ITT) population.) | 85
Not Completed | 1 | 1
Not completed — Administrative problems: | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cyclosporine A | Tacrolimus | Total
Number analyzed (Participants) | 84 | 85 | 169
Age Continuous [Mean (Standard Deviation); unit: Years] — Baseline measures are based on intention to treat (ITT) population.
  Years | 48.1 (12.069) | 49.9 (9.886) | 48.98 (11.029)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 30 | 61
  Male | 53 | 55 | 108

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Occurrence of Biopsy Proven Acute Rejection (BPAR) During the First 3 Months Post de Novo Liver Transplantation.
Description: A BPAR is defined when the investigator had a suspicion of an acute rejection, where the final clinical diagnosis confirmed the occurrence of an acute rejection, where a biopsy was performed that confirmed the presence of an acute rejection, and where anti-rejection treatment intervention was initiated. The efficacy measured the first rejections (clinically and biopsy proven rejections) at 3 months.
Time Frame: Month 3
Population: Intention to treat (ITT) population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Cyclosporine A | Tacrolimus
Number analyzed (Participants) | 84 | 85
Percentage of Participants | 33.3 | 32.9

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | Tacrolimus | Cyclosporine A
Serious Adverse Events (participants affected / at risk) | 42/86 | 33/85
Other Adverse Events (participants affected / at risk) | 84/86 | 85/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus (N=86) | Cyclosporine A (N=85)
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0
Megacolon (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Truncus coeliacus thrombosis (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0
Chest pain (General disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 11 | 4
Biliary dilatation (Hepatobiliary disorders) | 0 | 1
Biliary ischaemia (Hepatobiliary disorders) | 0 | 1
Biloma (Hepatobiliary disorders) | 2 | 0
Cholangitis (Hepatobiliary disorders) | 3 | 2
Cholestasis (Hepatobiliary disorders) | 0 | 2
Hepatic artery thrombosis (Hepatobiliary disorders) | 1 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic haemorrhage (Hepatobiliary disorders) | 1 | 0
Hepatic necrosis (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 1
Liver function test abnormal (Hepatobiliary disorders) | 1 | 0
Liver injury (Hepatobiliary disorders) | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 2 | 0
Graft versus host disease (Immune system disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Cytomegalovirus colitis (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 2 | 0
Hepatitis C (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 1
Septic shock (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Biliary anastomosis complication (Injury, poisoning and procedural complications) | 3 | 3
Hepatic haematoma (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Transplant failure (Injury, poisoning and procedural complications) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Amnesia (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1
Neurotoxicity (Nervous system disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 0
Nephropathy toxic (Renal and urinary disorders) | 0 | 2
Oliguria (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Brain hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis herpetiformis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Arterial haemorrhage (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1
Intra-abdominal haemorrhage (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus (N=86) | Cyclosporine A (N=85)
Anaemia (Blood and lymphatic system disorders) | 20 | 28
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 7
Cardiac failure (Cardiac disorders) | 5 | 4
Tachycardia (Cardiac disorders) | 5 | 7
Abdominal pain (Gastrointestinal disorders) | 14 | 24
Abdominal pain upper (Gastrointestinal disorders) | 10 | 9
Ascites (Gastrointestinal disorders) | 29 | 35
Constipation (Gastrointestinal disorders) | 26 | 32
Diarrhoea (Gastrointestinal disorders) | 26 | 54
Dyspepsia (Gastrointestinal disorders) | 4 | 5
Ileus (Gastrointestinal disorders) | 6 | 2
Impaired gastric emptying (Gastrointestinal disorders) | 2 | 7
Nausea (Gastrointestinal disorders) | 40 | 39
Vomiting (Gastrointestinal disorders) | 25 | 26
Chest pain (General disorders) | 7 | 3
Fatigue (General disorders) | 8 | 12
Oedema (General disorders) | 41 | 37
Pain (General disorders) | 8 | 10
Pyrexia (General disorders) | 25 | 33
Biloma (Hepatobiliary disorders) | 5 | 1
Cholestasis (Hepatobiliary disorders) | 4 | 8
Jaundice (Hepatobiliary disorders) | 6 | 0
- Unknown Infections - (Infections and infestations) | 23 | 18
Candidiasis (Infections and infestations) | 23 | 27
Clostridial infection (Infections and infestations) | 5 | 5
Cytomegalovirus infection (Infections and infestations) | 16 | 14
Enterobacter infection (Infections and infestations) | 12 | 9
Enterococcal infection (Infections and infestations) | 28 | 37
Epstein-Barr virus infection (Infections and infestations) | 2 | 7
Escherichia infection (Infections and infestations) | 27 | 19
Haemophilus infection (Infections and infestations) | 1 | 5
Herpes simplex (Infections and infestations) | 3 | 6
Infection (Infections and infestations) | 4 | 8
Pneumonia klebsiella (Infections and infestations) | 9 | 16
Pseudomonas infection (Infections and infestations) | 8 | 9
Staphylococcal infection (Infections and infestations) | 34 | 33
Streptococcal infection (Infections and infestations) | 8 | 9
Biliary anastomosis complication (Injury, poisoning and procedural complications) | 9 | 7
Procedural pain (Injury, poisoning and procedural complications) | 22 | 33
Diabetes mellitus (Metabolism and nutrition disorders) | 8 | 15
Fluid retention (Metabolism and nutrition disorders) | 8 | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 10
Hyperkalaemia (Metabolism and nutrition disorders) | 13 | 8
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 26
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 5
Dizziness (Nervous system disorders) | 8 | 12
Headache (Nervous system disorders) | 26 | 23
Paraesthesia (Nervous system disorders) | 13 | 7
Somnolence (Nervous system disorders) | 5 | 1
Tremor (Nervous system disorders) | 12 | 18
Anxiety (Psychiatric disorders) | 7 | 5
Delirium (Psychiatric disorders) | 9 | 5
Insomnia (Psychiatric disorders) | 30 | 46
Restlessness (Psychiatric disorders) | 10 | 15
Nephropathy toxic (Renal and urinary disorders) | 19 | 24
Oliguria (Renal and urinary disorders) | 5 | 7
Polyuria (Renal and urinary disorders) | 16 | 10
Renal failure (Renal and urinary disorders) | 5 | 4
Renal impairment (Renal and urinary disorders) | 7 | 12
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 16
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 24 | 21
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 12
Rash (Skin and subcutaneous tissue disorders) | 6 | 5
Hypertension (Vascular disorders) | 33 | 21
Hypotension (Vascular disorders) | 7 | 6
Intra-abdominal haemorrhage (Vascular disorders) | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.